CLINICAL TRIAL: NCT03837249
Title: Self-Management of Sleep Among Older Adults Using Personal Monitoring: A Feasibility Study
Brief Title: Self-Management of Sleep Among Older Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Responsible Party: Principal Investigator, Raeann G LeBlanc, Assistant Clinical Professor, University of Massachusetts, Amherst
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2018-5225
Record Dates: First submitted 2019-01-24; First posted 2019-02-12 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Sleep Disturbance
Keywords: Older People; Sleep Disturbance; Self-Monitoring; Self-Management; Social Support; Wrist-worn Actigraphy
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Intervention Model Description: Comparative control - 3 group
Who Masked: Participant
Masking Description: One group - personal sleep monitoring data with-held then provided after the intervention period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Passive Personal Sleep Monitoring (Placebo Comparator): Wears personal sleep monitor but does not actively self-monitor (will have access to the sleep data and self-monitoring after 4 weeks).
  Interventions: Device: Personal Sleep Monitoring
- Individual Personal Sleep Monitoring (Active Comparator): Wears personal sleep monitor and actively self-monitoring sleep and using data to self-manage sleep.
  Interventions: Device: Personal Sleep Monitoring
- Socially Supported Sleep Monitoring (Active Comparator): Wears a personal sleep monitor, actively self-monitoring using sleep data to self-manage sleep and shares data for supportive self-management.
  Interventions: Device: Personal Sleep Monitoring

INTERVENTIONS:
Device: Personal Sleep Monitoring — Wearable Sleep Self-Monitoring Device (Actigraphy)
  Other Names: Personal Sleep Monitor

SUMMARY:
The purpose of this study is to test the feasibility of older persons use of a personal sleep monitoring device(PSMD)to improve self-management of sleep. Disrupted sleep occurs in up to 50% of persons over the age of 65 with chronic health conditions. Impaired sleep negatively influences subjective and objective health outcomes.To improve their sleep, older adults with chronic health conditions could benefit from objective information, available through personal health monitoring devices, about their current and changing sleep patterns. Based on this information, sleep self-management interventions can be individualized and shared, and associations between sleep and health changes may be better managed.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* Self-report difficulty sleeping
* Willingness to wear the PSMD for four weeks
* Cognitive abilities (Mini Cog of 5 or above).

Exclusion Criteria:

* Under the age of 65
* Presence of known sleep disorders
* Severe cognitive or neurosensory impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Use of A Personal Sleep Monitoring Device (PSMD) | up to 4 weeks
  Demonstrates use of Personal Sleep Self-Monitor through data downloads and self-report
Changes in Sleep | Week 1 and Week 4
  Demonstrated sleep changes indicated by change in BRCS NINR PROMIS SF V1 Sleep Disturbance Scale 6a (a 6 item, 5 point likert scale with higher scores reflecting more sleep disturbance and lower scores less.
Changes in Health | Week 1 and Week 4
  Demonstrated health changes indicated by change in BRCS NINR PROMIS Global Health Short Form Scale 10a (10 item, 5 point likert scale) with higher scores reflecting better health (3 items reverse scoring)

SECONDARY OUTCOMES:
Usability of PSMD | Week 2 and 4
  Demonstrated through adapted System Usability Scale Scores (10 items, 5 point likert scale) with high agreement demonstrating higher levels of satisfaction using the device

CONTACTS AND LOCATIONS:
Overall Officials: Raeann G LeBlanc, PhD, DNP, Principal Investigator — University of Massachusetts, Amherst
Locations (1):
- University of Massachusetts, Amherst, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
IPD data will be shared de-identified as a GUID with the cdRNS data base.